CLINICAL TRIAL: NCT00401440
Title: Comparison of Twq Different Regimen of Vaginal Misoprostol for Nid Trimester MTP
Brief Title: Comparison of Two Regimens of Misoprostol for Second Trimester Medical Termination of Pregnancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nilratan Sircar Medical College (Other Government)
Responsible Party: Chairperson , I Ethical Committee & Principal, Nilratan Sircar Medical College , Kolkata
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3-Chaudhuri
Record Dates: First submitted 2006-11-16; First posted 2006-11-20 (Estimated); Last update posted 2010-03-12 (Estimated); Status verified 2008-12

CONDITIONS: Induced Abortion
Keywords: Medical termination of pregnancy; Induction of abortion; Misoprostol; MTP in second trimester; 400 microgram vaginal misoprostol
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): 400 microgram vaginal misoprostol tablet will be applied every 6 hours with a maximum of 4 doses
  Interventions: Drug: Misoprostol
- B (Active Comparator): 400 microgram vaginal misoprostol tablet will be applied every 12 hours with a maximum of 4 doses
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — 400 microgram vaginal misoprostol tablet will be applied every 6 hours with a maximum of 4 doses
  Arms: A
Drug: Misoprostol — 400 microgram vaginal misoprostol tablet will be applied every 12 hours with a maximum of 4 doses
  Arms: B

SUMMARY:
The hypothesis of the study is that the induction abortion interval time will be significantly shorter in the group receiving vaginal misoprostol every six hours in comparison to the group who are receiving vaginal misoprostol every twelve hours.

DETAILED DESCRIPTION:
Objectives:

Misoprostol, a prostaglandin analogue, is principally used to prevent peptic ulcer disease induced by nonsteroidal anti-inflammatory agents .It has been shown to induce second trimester abortion .However , the optimal regimen has not been determined .Studies have used doses ranging 200- 800 microgram misoprostol at interval ranging from 3-12 hours.1,2,3,4,5 In our previous study we have compared intravaginal misoprostol with extra amniotic ethacridine lactate for second trimester MTP.6 In this study we have observed that misoprostol is highly effective( success rate 95%) for second trimester MTP with minimal side effects .& intravaginal misoprostol results in significantly shorter induction abortion interval in comparison to extra amniotic ethacridine lactate .Induction abortion interval in this study for misoprostol was 15.5 hours and the dosage of misoprostol was 400 microgram vaginally every 12 hours with a maximum of 4 doses .Success rate and induction abortion interval are the major factors of clinical importance for second trimester MTP . Our aim is to establish a dosage schedule of misoprostol which will result in high success rate in mid trimester MTP with further shortening of induction abortion interval Our study hypothesis is that using 400 microgram of vaginal misoprostol at six hour interval will result in significant shortening of induction abortion interval in comparison to 400 microgram vaginal misoprostol at 12 hour interval.

Methods - A prospective randomized comparative clinical trial will be conducted over 200 women.

Women attending the hospital for mid trimester MTP i.e. 12-20 weeks of pregnancy will be taken up for the study. Gestational age will be determined from LMP & per abdominal findings. Ultrasonography will be done in selected women where clinical finding is unreliable . All women will be examined for vital parameters and routine hematological and urine examination will be done. Randomization will be done using a table of random numbers .A written consent for inclusion in the study will be taken from all patients who will be included in the study.

In one group women will receive 400 microgram vaginal misoprostol tablet at interval of 12 hours with a maximum of four doses.

In other group women will receive 400 microgram vaginal misoprostol tablet at an interval of 6 hours with a maximum of four doses.

Failure of procedure in both groups will be defined as failed expulsion of fetus at 48 hours or as the occurrence of systemic adverse signs and symptoms severe enough to preclude the use of additional drugs.

The patient's vital signs will be monitored every four hours and the occurrence of signs and symptoms, such as fever, pain, vomiting, and diarrhea will be recorded. After expulsion of the fetus and placenta, check curettage will be done in every case. Completeness of abortion will be defined as expulsion of both placenta and fetus without operative assistance. The induction abortion interval will be defined as time from administration of 1st dose of Misoprostol to abortion of fetus. Hemorrhage will be defined as an estimated blood loss exceeding 500 ml or need to blood transfusion. Fever will be defined as rise of temperature 100.4˚ F or more occurring 24 hours or more after pregnancy termination.

The following parameters will be studied (1) Induction abortion interval (2) Completeness of procedure (3) Failure of abortion (4) side effects (5) cost per procedure.

Statistical analysis will be carried out with Epi Info statistical software.

ELIGIBILITY:
Inclusion Criteria:

* Women fulfilling indications of Medical Termination Of Pregnancy Act of India
* 12-20 weeks of pregnancy

Exclusion Criteria:

* Women with previous uterine surgery
* Contraindication of misoprostol use

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 185 (Actual)
Dates: Start 2007-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
induction abortion interval | 48 hours

SECONDARY OUTCOMES:
Success rate | 48 hours
Side effects | 48 hours
complete expulsion of products of conception | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Snehamay Chaudhuri, MBBS,MD,DNB, Principal Investigator — Nilratan Sircar Medical College , 138,AJC Bose Road , Kolkata,700014,West Bengal , India.
Locations (1):
- Department of Gynae & Obstetrics, Nilratan Sircar Medical College , Kolkata, Kolkata, West Bengal, India

REFERENCES:
- See also: A comparison of intra vaginal misoprostol with extra amniotic ethacridine lactate for second trimester MTP, J Obstet Gynecol India .56.6:2006.518-521 — http://medind.nic.in/jaq/t06/i6/jaqt06i6p518.pdf